CLINICAL TRIAL: NCT00282269
Title: Pilot Study of Early and Prolonged Hypothermia in Severe Traumatic Brain Injury in Children
Brief Title: Hypothermia in Traumatic Brain Injury in Children (HiTBIC)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Australia and New Zealand Intensive Care Society (Other)
Responsible Party: Dr Michael Yung, Chair, Paediatric Study Group, Clinical Trials Group, ANZICS
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: NTX/06/02/002
Record Dates: First submitted 2006-01-25; First posted 2006-01-26 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2009-06

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; Children; Hypothermia; Outcome; Intensive Care; Magnetic resonance Imaging
MeSH Terms: conditions — Brain Injuries, Traumatic; Hypothermia | interventions — Hypothermia, Induced

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Induced Hypothermia — Induced Hypothermia within 6 hours of injury and maintained for a minimum of 72 hours

SUMMARY:
The purpose of this study is:

* To determine the safety and feasibility of performing an international multi-centre randomized control trial of early and prolonged hypothermia to improve outcome in children with severe traumatic brain injury (TBI).
* To determine whether in children with severe traumatic brain injury, prolonged initial hypothermia (minimum 72 hours at 32-33 degrees) improves the proportion of good outcomes 12 months after injury when compared to initial normothermia (36-37 degrees).

DETAILED DESCRIPTION:
We propose to do a pilot study of 50 children admitted with severe TBI to paediatric intensive care units in Australia and New Zealand. Severe TBI will be defined as children with either (i) Glasgow Coma Scale (GCS) ≤ 8 and an abnormal CT scan or (ii) motor score of ≤ 3 and normal CT scan. Children will be included only if they can be randomised within 6 hours of the injury occurring. Patients will be stratified a priori by (i) centre and (ii) Glasgow Coma Score. One half will be cooled to 32-33°C for 72 hours and then slowly rewarmed. If intracranial hypertension occurs during or after rewarming, the hypothermia group will have cooling continued until intracranial pressure (ICP) is controlled. The other half will have their temperature maintained at 36-37°C. All other aspects of care will be managed with a standardised protocol.

The purpose of this pilot study is to establish the feasibility of doing an outcome study with other international centres. It will also assess the safety of more prolonged cooling and protocol adherence. Primary outcomes will be the frequency of adverse events related to hypothermia, recruitment rates and protocol adherence. These children may also be able to be included in a larger trial.

The primary aim of the outcome study will be to determine whether, in children with severe TBI, prolonged initial hypothermia improves the proportion with good outcome 12 months after injury when compared to initial normothermia. Outcome will be assessed at 6 and 12 months. The primary outcome measure will be a Paediatric Cerebral Performance Category (PCPC) at 12 months after the date of injury, dichotomized to poor outcome (categories 4-6) and good outcome (categories 1-3). Secondary outcome measures will be (i) PCPC at 6 after injury (ii) standardised tests (intelligence and memory, functional outcome, attention, executive functions) 12 months after injury (iii) ICP and cerebral perfusion pressure (CPP) during the first 5 days of treatment (v) frequency and nature of interventions to control ICP/CPP (vi) duration of mechanical ventilation and (vii) potential adverse events.

ELIGIBILITY:
Inclusion Criteria:

* have a severe traumatic brain injury as defined by either a GCS ≤ 8 and an abnormal CT scan (intracranial hemorrhage, cerebral edema or diffuse axonal injury) or a motor score ≤ 3 and normal CT scan
* are aged between 1 and 16 years
* are mechanically ventilated

Exclusion Criteria:

* are not randomized by 6 hours after injury
* have penetrating brain injuries
* have fixed dilated pupils and GCS = 3
* have proven cervical spinal cord injury
* have more than mild neurodevelopmental disability prior to injury
* have an acute isolated epidural hematoma and are expected to recover rapidly after surgical removal
* have had a post-traumatic seizure with a normal CT scan
* have refractory shock, defined as systolic blood pressure more than 2 standard deviations (SD) below the mean for age despite 80ml/kg intravenous fluid resuscitation

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2006-11; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Paediatric Cerebral Performance Category (PCPC) at 12 months after injury | 12 months
Recruitment Rates | Recruitment completion
Adverse Events | Recruitment completion

SECONDARY OUTCOMES:
Intracranial pressure(ICP)/Cerebral perfusion pressure(CPP) control | Recruitment completion
Duration of mechanical ventilation | Recruitment completion
Intensive care and hospital length of stay | Recruitment completion
Neuropsychological Outcome | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: John Beca, FJFICM, Principal Investigator — Starship Children's Hospital, Auckland, New Zealand
Locations (7):
- Australia (6):
  - Royal Alexandra Hospital for Children, Sydney, New South Wales
  - Sydney Children's Hospital, Sydney, New South Wales
  - Queensland Paediatric Intensive Care Services, Brisbane, Queensland
  - Women's and Children's Hospital, Adelaide, South Australia
  - Royal Children's Hospital, Melbourne, Victoria
  - Princess Margaret Hospital, Perth, Western Australia
- Starship Children's Hospital, Auckland, New Zealand